CLINICAL TRIAL: NCT00070213
Title: Drug Treatment for Bowel Cancer: Making the Best Choices When a Milder Treatment is Needed
Brief Title: Leucovorin and Fluorouracil With or Without Oxaliplatin Compared to Capecitabine With or Without Oxaliplatin in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Cheryl Pugh, Clinical Project manager for FOCUS2 for Sponsor, Medical Research Council
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000330142; NCRI-FOCUS2; MRC-CR09; EU-20303
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV rectal cancer; stage IV colon cancer; recurrent rectal cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MdG (modified de Gramont) (Active Comparator): 2 weekly 5FU/FA schedule
  Interventions: Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Procedure: quality-of-life assessment
- OxMdG (80%) for 12 weeks (Experimental): MdG + oxaliplatin
  Interventions: Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: quality-of-life assessment
- Capcitabine (Experimental)
  Interventions: Drug: capecitabine; Procedure: quality-of-life assessment
- OxCap (Experimental)
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: FOLFOX regimen
  Arms: MdG (modified de Gramont); OxMdG (80%) for 12 weeks
Drug: capecitabine
  Arms: Capcitabine; OxCap
Drug: fluorouracil
  Arms: MdG (modified de Gramont); OxMdG (80%) for 12 weeks
Drug: leucovorin calcium
  Arms: MdG (modified de Gramont); OxMdG (80%) for 12 weeks
Drug: oxaliplatin
  Arms: OxCap; OxMdG (80%) for 12 weeks
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as leucovorin, fluorouracil, capecitabine, and oxaliplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether leucovorin and fluorouracil with or without oxaliplatin is more effective than capecitabine with or without oxaliplatin in treating patients who have metastatic colorectal cancer.

PURPOSE: This randomized phase III trial is studying four different chemotherapy regimens to compare how well they work in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with metastatic colorectal adenocarcinoma treated with leucovorin calcium and fluorouracil with vs without oxaliplatin or capecitabine with vs without oxaliplatin.
* Compare the quality of life of patients treated with these fluorouracil-based vs capecitabine-based regimens.

Secondary

* Compare the failure-free and overall survival of patients treated with these regimens.
* Compare the toxic effects and adverse events associated with these regimens in these patients.
* Compare the limited health assessments of patients treated with these regimens.
* Compare the health economics associated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 4 treatment arms and receive 12 weeks of therapy.

* Arm I (MdG regimen): Patients receive leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression during or within 8 weeks of the completion of this regimen may cross over and receive second-line therapy on arm II.

* Arm II (OxMdG regimen): Patients receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression during or within 8 weeks of the completion of this regimen may receive second-line therapy or supportive care off-study.

* Arm III (Cap regimen): Patients receive oral capecitabine twice daily on days 1-15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression during or within 8 weeks of the completion of this regimen may cross over and receive second-line therapy on arm IV.

* Arm IV (OxCap regimen): Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression during or within 8 weeks of the completion of this regimen may receive second-line therapy or supportive care off-study.

All patients are then re-evaluated at least every 6 weeks and begin another 12 weeks of therapy at any evidence (e.g., clinical, radiological, or tumor marker) of disease progression. Patients with chemo-sensitive disease may repeat alternating 12-week therapy sessions and evaluation periods indefinitely.

Quality of life is assessed at baseline, at 12-14 weeks, at 24 weeks, and then every 3 months thereafter.

Patients are followed every 3 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 460 patients (115 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma, defined by 1 of the following:

  * Prior or current histologically confirmed primary adenocarcinoma of the colon or rectum with clinical/radiological evidence of advanced/metastatic disease
  * Histologically or cytologically confirmed metastatic adenocarcinoma with clinical/radiological evidence of colorectal primary tumor
* Unidimensionally measurable disease
* Unfit and unsuitable for full-dose combination chemotherapy, which would include 1 of the following circumstances:

  * Unsuitable or unwilling to be entered into any full-dose chemotherapy protocol
  * Ineligible or unsuitable for first-line standard combination as per National Institute of Clinical Excellence guidance

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN

Renal

* Creatinine clearance greater than 50 mL/min OR
* Glomerular filtration rate greater than 30 mL/min

Cardiovascular

* No uncontrolled angina
* No recent myocardial infarction

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No partial or complete bowel obstruction
* No concurrent severe uncontrolled medical illness that would preclude study treatment
* No psychiatric or neurological condition that would preclude giving informed consent or complying with oral study medication
* No other prior or concurrent malignant disease that would preclude study treatment or assessment of response
* No prior neuropathy greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 months since prior adjuvant chemotherapy with fluorouracil with or without leucovorin calcium
* More than 1 month since prior rectal chemoradiotherapy with fluorouracil with or without leucovorin calcium
* No prior systemic palliative chemotherapy for metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy

Surgery

* Not specified

Other

* No concurrent brivudine or sorivudine

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2003-09; Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
Compare progression-free survival (PFS) in pts. treated w/ leucovorin calcium + fluorouracil (MdG) vs leucovorin calcium + fluorouracil + oxaliplatin (OxMdG) and in pts. treated w/ capecitabine (Cap) vs capecitabine + oxaliplatin (OxCap) at 1 yr | PFS
  Compare progression-free survival (PFS) in pts. treated w/ leucovorin calcium + fluorouracil (MdG) vs leucovorin calcium + fluorouracil + oxaliplatin (OxMdG) and in pts. treated w/ capecitabine (Cap) vs capecitabine + oxaliplatin (OxCap) at 1 yr
Compare health assessment in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap at baseline and 14 weeks | Baseline and 14 weeks
  Compare health assessment in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap at baseline and 14 weeks

SECONDARY OUTCOMES:
Compare health assessment, including quality of life, in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap at baseline and 14 and 24 weeks | Baseline, 14 and 24 weeks
  Compare health assessment, including quality of life, in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap at baseline and 14 and 24 weeks
Compare toxicity/adverse events in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap | post 24 weeks
  Compare toxicity/adverse events in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap
Compare overall failure-free survival in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap | post 24 weeks
  Compare overall failure-free survival in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap
Compare overall survival in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap | post 24 weeks
  Compare overall survival in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap
Compare health economics in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap | Baseline, 14 and 24 weeks
  Compare health economics in patients treated with MdG vs OxMdG and in patients treated with Cap vs OxCap
Compare health assessment in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap | Baseline, 14 and 24 weeks
Compare toxicity/adverse events in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap at baseline and 24 weeks | Baseline and 24 weeks
  Compare toxicity/adverse events in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap at baseline and 24 weeks
Compare patients acceptability in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap | post 24 weeks
  Compare patients acceptability in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap
Compare PFS in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap | post 24 weeks
  Compare PFS in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap
Compare health economics in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap | Baseline, 14 and 24 weeks
  Compare health economics in patients treated with MdG vs Cap and in patients treated with OxMdG vs OxCap

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Seymour, MA, MD, FRCP, Principal Investigator — Cookridge Hospital; Gareth Griffiths, Study Chair — Medical Research Council
Locations (4):
- United Kingdom (4):
  - Cookridge Hospital, Leeds, England
  - Clinical Trials and Research Unit of the University of Leeds, Leeds, England
  - Medical Research Council Clinical Trials Unit, London, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Seymour MT, Thompson LC, Wasan HS, Middleton G, Brewster AE, Shepherd SF, O'Mahony MS, Maughan TS, Parmar M, Langley RE; FOCUS2 Investigators; National Cancer Research Institute Colorectal Cancer Clinical Studies Group. Chemotherapy options in elderly and frail patients with metastatic colorectal cancer (MRC FOCUS2): an open-label, randomised factorial trial. Lancet. 2011 May 21;377(9779):1749-59. doi: 10.1016/S0140-6736(11)60399-1. Epub 2011 May 11. PMID 21570111
- [Result] Seymour MT, Maughan TS, Wasan HS, et al.: Capecitabine (Cap) and oxaliplatin (Ox) in elderly and/or frail patients with metastatic colorectal cancer: the FOCUS2 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-9030, 500s, 2007.
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://events.cancer.gov/sites/default/files/assets/DCP-olderadultaccrual/Study%20Design%20and%20Assessment.pdf